CLINICAL TRIAL: NCT04017715
Title: Effects of Cricket Injury Prevention Program on National Cricket Players of Rawalpinidi
Brief Title: Effect of Injury Prevention Program on Cricketers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC/00510 Amna Imran
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Sports Physical Therapy
Keywords: cricket injury prevention program,sports injuries,
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- warm up (Experimental): warm up exercises
  Interventions: Other: Experimental: warm up
- cool down (Experimental): cool down exercises
  Interventions: Other: Experimental: cool down
- control (Active Comparator): Following conventional protocol
  Interventions: Other: No intervention: control

INTERVENTIONS:
Other: Experimental: warm up — Phase 1 is dynamic stretching and running exercises which includes, A jogging ,B walking lunge and sweeps, C hip in and out running : jog 3 steps stop and do "hip in"/hip out" for Phase 2 is strength and agility which includes A- squat, B- push-ups: wide palmer push-ups. C vertical jumps. D- lateral jump. E- nordic hamstrings,. F (a)- shoulder external rotations, F(b)- modified inverted rows, Phase 3 is balance and core strength which includes A- modified ankle discs, B - planks: standard forward planks 2 repetitions for 30secs. C- side planks: standard side planks on both sides 1 repetition for 20 secs. Da- bird-dog,Db- modified back extensions, Phase 4 is run sprint which includes A- run sprint: 100% speed running between running (20m) with 1 repetition
  Arms: warm up
Other: Experimental: cool down — Phase 1 is dynamic stretching and running exercises which includes, A jogging ,B walking lunge and sweeps, C hip in and out running : jog 3 steps stop and do "hip in"/hip out" for Phase 2 is strength and agility which includes A- squat, B- push-ups: wide palmer push-ups. C vertical jumps. D- lateral jump. E- nordic hamstrings,. F (a)- shoulder external rotations, F(b)- modified inverted rows, Phase 3 is balance and core strength which includes A- modified ankle discs, B - planks: standard forward planks 2 repetitions for 30secs. C- side planks: standard side planks on both sides 1 repetition for 20 secs. Da- bird-dog,Db- modified back extensions, Phase 4 is run sprint which includes A- run sprint: 100% speed running between running (20m) with 1 repetition
  Arms: cool down
Other: No intervention: control — sprint exercise and general stretching as conventional protocol as follows in star club
  Arms: control

SUMMARY:
The main aim of the study is to prevent the injuries during cricket.Total 60 players were included in the study. 20 players were in warm up group,20 players were in cool down group and 20 players in control group.Base line assessment was by 100m sprint, Illinios agility test, 3 minute burpee test, SEBT and plank. After intervention of 6 weeks assessment will be done again by using the same tests.

DETAILED DESCRIPTION:
Cricket is referred to as the second most popular game in world after football and in subcontinent along with south east Asian countries its popularity is increasing day by day it's also referred to as gentle's man game and was regarded as relatively injury free, but recently all witnessed that, changes brought to the cricketing world thus making the game more exciting for the viewers and demanding for players , as a result of these changes and high frequency of matches the game of cricket is no longer an injury free and involves risk of moderate to high level of injuries. These changes in game posed their effects on the players and now they are required to have and maintain high level of fitness In addition to technical skill, however this fitness regimen is also causing problems for players i.e. making them prone to overuse injuries a survey conducted by BSC and ACB reported 2.6 injuries and 24.2 injuries per 10,000 players hours respectively and there are studies to prove that most injury cases are reported in specific stages of the season. The major areas of concern are impact injuries to the head, face and fingers and injuries to the back.

Here it's worth defining that what actually is a injury An injury, which could be an acute or an overuse injury, is defined as any physical damage that took place during a game play, practice or training session and which prevented the player from completing that particular game, practice or training session. In similar way a cricket injury is defined as harmful condition or other medical related issue faced by the player that inhibits him/her from being selected for play or makes the player unable to resume his/her normal game for a partial or whole game when required by either the rules or the team captain.The most common injuries reported are hamstring strains, side strains, groin injuries, wrist and hand injuries, and lumbar soft tissue injuries .

While all cricketers are at the a risk of assuming an acute soft tissue injury to lower limb along the Fast bowlers fall under the highest risk category, as well as role-specific injuries. According to statistical data presented by Stretch & Venter 66% of overall reported injuries fall in serious category, while chronic and acute-on-chronic made up 12% and 22%, respectively. Where reported Soft-tissue injuries were primarily muscle related injuries constituting up to (41%).

According to Stretch The frequency of injury to the head, neck, and face varied from 5.4% to 25%, and the upper limbs accounted for 19.8% to 34.1% of injuries. Back and trunk injuries accounted for 18.0% to 33.3% of the injuries, and lower-limb injuries accounted for 22.8% to 50.0%. Most were first-time injuries; recurrent injuries from the previous season accounted for 23.9% to 29.8%, and injuries sustained during the season recurring again during the same season, 22.7% to 36.8%. Dhillon et al., report that upper limb injuries are more common in cricket players and account for 16.8%

Dhillon et al., in their research also report that 62.5% injuries were severe enough to prevent cricketers from returning to play for more than 4 weeks. Orchard et al gave a further insight to Injury prevalence (the percentage of players missing due to an injury at any given time) was 14% for pace bowlers, 4% for spin bowlers, 4% for batsmen, and 2% for wicket keeper.

In researches carried out by Dhillon et al, the percentage of injuries reported for fast bowlers as compared to rest is quite high this is due to the fact that pace bowling involves repetitive twisting, extension and rotation of trunk and at the same time bowlers are absorbing high reaction forces over a short period of time. These movements, if performed incorrectly or too frequently, can lead to overuse injuries of the back, particularly in elite and high-level cricketers

An increased throwing workload is a risk factor for the development of upper limb injury in elite cricketers.Stretch & Venter conducted a longitudinal study showing a pattern for the causes of injuries sustained by the cricketers and reported that the young fast bowlers are most likely to sustain an acute soft tissue injury to the lower limb in early part of the cricketing season while playing in games of cricket or practice sessions. Cross-sectional studies have also demonstrated that spinal overuse injuries occur more frequently to cricketers adopting a mixed bowling action than to those who favor a front or a side-on bowling technique

Strategies are placed in order to ensure that cricketers do not adopt the mixed action or bowl too fast for extended periods thus helping to prevent the back injuries. Along with injuries resulting from impacts, injuries from cricket ball impact can also occur and are more common during low level competition or informal participation. Because of the potential severity of these impacts, a range of protective equipment ranging from body padding to gloves and face protectors are now common features of standard cricket equipment. Although a number of measures to prevent cricket injuries have been widely suggested in the literature, there have been very few studies that have formally assessed their effectiveness in preventing injury. Further research is needed to gain a greater understanding of the bio mechanics of cricket actions, the mechanisms of resultant injuries and the role of various risk factors in injury causation. The extent of the sports injury problem must be identified and described. Secondly the factors and mechanisms which play a part in the occurrence of sports injuries have to be identified. The third step is to introduce measures that are likely to reduce the future risk and/or severity of sports injuries.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16-30 years
* Male cricketers registered with PCB
* Players attending minimum three sessions per week

Exclusion Criteria:

* Players having any of the following :
* neuromusculoskeletal ,
* cardiovascular, or systematic pathology.

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — only male participants were included as per availibility
Enrollment: 55 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
3 minute burpee test | 6th week
  changes from the baseline, The three MBT can be used with authenticity in order to judge endurance & strength capabilities amid young women. The "training trend" has to be abolished prior to conducting the test that is used for assessment of endurance-strength abilities. A minimum of 5 repeats must be executed for the test to provided results. time will be noted in seconds
Illinois Agility Run Test: | 6th week
  changes from the baseline, Agility is acrucial module of any team sports, however it is not continuously and normally tested, due to the fact its quite challenging to interpret its results. The Illinois Agility Test is a generally used as a test of nimbleness in sportsperson and per se there are several norms available.This is a modest test to govern, requiring little equipment this test also tests out the player's capacity to turn in altered directions and unlike angles. time will be noted in seconds
Plank test: | 6th week
  changes from the baseline, The plank test is a general test carried out to measure core strength also can be utilized as a fitness drill for enhancing core strength. Purpose of this test is to measure the control and endurance of the back/core stabilizing muscles.time will be noted in seconds
SEBT | 6th week
  changes from the baseline, The "Star Excursion Balance Test" or "SEBT"is a vigorous test that involves strength, flexibility, and proprioception.
  The SEBT can also be used to compare balance ability among different sports and to assess physical performance. Research suggests to use this test as a screening tool for sport participation as well as a post-rehabilitation test to ensure dynamic functional symmetry. It has also been shown that the performance of SEBT improves after training. time will be noted in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Faheem Afzal, MSSPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maquirriain J, Ghisi JP. Uncommon abdominal muscle injury in a tennis player: internal oblique strain. Br J Sports Med. 2006 May;40(5):462-3. doi: 10.1136/bjsm.2005.023457. PMID 16632581
- [Background] Heiser TM, Weber J, Sullivan G, Clare P, Jacobs RR. Prophylaxis and management of hamstring muscle injuries in intercollegiate football players. Am J Sports Med. 1984 Sep-Oct;12(5):368-70. doi: 10.1177/036354658401200506. PMID 6496833
- [Background] Drezner JA. Practical management: hamstring muscle injuries. Clin J Sport Med. 2003 Jan;13(1):48-52. doi: 10.1097/00042752-200301000-00009. No abstract available. PMID 12544164
- [Background] Worrell TW. Factors associated with hamstring injuries. An approach to treatment and preventative measures. Sports Med. 1994 May;17(5):338-45. doi: 10.2165/00007256-199417050-00006. PMID 8052770
- [Background] Morton S, Barton CJ, Rice S, Morrissey D. Risk factors and successful interventions for cricket-related low back pain: a systematic review. Br J Sports Med. 2014 Apr;48(8):685-91. doi: 10.1136/bjsports-2012-091782. Epub 2013 May 10. PMID 23666021
- [Background] Merlino J, Perisa J. Low back pain in a competitive cricket athlete. Int J Sports Phys Ther. 2012 Feb;7(1):101-8. PMID 22319683
- [Background] Nealon AR, Kountouris A, Cook JL. Side strain in sport: a narrative review of pathomechanics, diagnosis, imaging and management for the clinician. J Sci Med Sport. 2017 Mar;20(3):261-266. doi: 10.1016/j.jsams.2016.08.016. Epub 2016 Aug 28. PMID 27616432